CLINICAL TRIAL: NCT07259109
Title: Psychotherapy and Psychopathology in Adolescence: an Observational Study
Brief Title: Psychopathology in Adolescence
Status: Enrolling by invitation | Type: Observational
Sponsor: IRCCS Centro Neurolesi Bonino Pulejo (Other)
Responsible Party: Sponsor
Other Study IDs: PSY25
Record Dates: First submitted 2025-07-04; First posted 2025-12-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-07

CONDITIONS: Anxiety Disorders; Depressive Disorder; Obsessive-Compulsive Disorder; Mental Health; Adolescent - Emotional Problem; Psychoterapy
MeSH Terms: conditions — Anxiety Disorders; Depressive Disorder; Obsessive-Compulsive Disorder; Psychological Well-Being

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- CBT Group: Participants receiving Cognitive Behavioral Therapy (CBT) as part of routine clinical care for adolescent psychopathology.
- BST Group: Participants receiving Brief Strategic Therapy (BST) as part of routine clinical care for adolescent psychopathology.

SUMMARY:
This observational study aims to evaluate the effectiveness of two different psychotherapy approaches-Cognitive Behavioral Therapy (CBT) and Brief Strategic Therapy (BST)-in treating adolescents with psychological disorders. The study will follow adolescents aged 12 to 20 who are receiving psychotherapy as part of their routine clinical care at the IRCCS Centro Neurolesi "Bonino-Pulejo" in Messina, Italy. Participants will not be randomly assigned to a treatment; instead, their natural clinical path will be observed. Data will be collected through standardized psychological assessments at the beginning, during, and after the therapy, as well as at follow-ups at 3 and 9 months. The goal is to understand which therapeutic model is more effective in improving symptoms, quality of life, and self-esteem in adolescents, and how individual and family factors influence treatment outcomes.

DETAILED DESCRIPTION:
This is a 5-year observational study evaluating the effectiveness and clinical characteristics of two psychotherapy approaches-Cognitive Behavioral Therapy (CBT) and Brief Strategic Therapy (BST)-in adolescents with psychiatric disorders. Patients aged 12 to 20 receiving care at the IRCCS Centro Neurolesi "Bonino-Pulejo" will be followed according to standard clinical practice, without random assignment. Psychopathological symptoms, self-esteem, and quality of life will be assessed at multiple time points (baseline, mid-treatment, end of treatment, and 3- and 9-month follow-ups) using standardized psychological tools. A propensity score matching method will be applied to reduce selection bias between treatment groups. The study also aims to identify predictors of treatment response and explore the influence of clinical and family-related factors on therapeutic outcomes. Data will be analyzed using both intra-group and inter-group statistical comparisons.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents aged 12 to 20 years
* Clinical diagnosis of a psychiatric disorder according to DSM-5 criteria
* Intelligence Quotient (IQ) ≥ 80
* Written informed consent signed by participant and/or legal guardian

Exclusion Criteria:

* Comorbid diagnosis of major neuropsychiatric disorders (e.g., autism spectrum disorder, schizophrenia)
* Intelligence Quotient (IQ) ≤ 79
* Lack of signed informed consent

Ages: 12 Years to 20 Years | Sex: All
Age Groups: Child, Adult
Study Population: Adolescents aged 12 to 20 years with clinically diagnosed psychiatric disorders, referred to the Child and Adolescent Psychiatry Unit at IRCCS Centro Neurolesi "Bonino-Pulejo" in Messina, Italy. All participants will be receiving psychotherapy (CBT or BST) as part of standard clinical care.
Sampling Method: Non-Probability Sample
Enrollment: 192 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2030-12 (Estimated); Study Completion 2031-03 (Estimated)

PRIMARY OUTCOMES:
Child Behavior Checklist (CBCL) | Baseline, Month 3, Month 6, Month 9, and Month 12
  The Child Behavior Checklist (CBCL) is a standardized parent-report questionnaire used to assess a wide range of emotional and behavioral problems in children. Higher scores indicate greater levels of emotional and behavioral difficulties.
SAFA General Screening Scales | Baseline, Month 3, Month 6, Month 9, and Month 12
  The SAFA (Self Administrated Psychiatric Scales for Youths and Adolescents) is a comprehensive set of standardized self-report questionnaires used to assess emotional and psychiatric symptoms in children and adolescents aged 8 to 18 years. The full battery includes six scales:
  * SAFA-A (Anxiety)
  * SAFA-D (Depression)
  * SAFA-O (Obsessive-Compulsive Symptoms)
  * SAFA-S (Somatic Complaints)
  * SAFA-P (Psychogenic Psychotic Symptoms)
  * SAFA-F (Eating Disorders)
  Each scale produces a raw score, which is then converted into a standardized score. Total scores for each domain range approximately from 0 to 100, although precise ranges vary slightly by scale and age group. Higher scores reflect more severe emotional or psychological difficulties, i.e., a worse outcome.
Personality Inventory for DSM (PID) | Baseline, Month 3, Month 6, Month 9, and Month 12
  The Personality Inventory for DSM-5 (PID-5) is a standardized self-report instrument developed to assess maladaptive personality traits aligned with the DSM-5 alternative model for personality disorders. It includes 220 items, rated on a 4-point Likert scale (0 = Very False or Often False; 3 = Very True or Often True), and provides scores on five broad domains:
  * Negative Affectivity
  * Detachment
  * Antagonism
  * Disinhibition
  * Psychoticism
  Scores range from 0 to 660 (sum of all item scores), although domain and facet scores are typically reported separately. Higher scores reflect more severe or dysfunctional personality traits (i.e., a worse outcome).
Columbia-Suicide Severity Rating Scale (C-SSRS) | Baseline, Month 3, Month 6, Month 9, and Month 12
  The Columbia-Suicide Severity Rating Scale (C-SSRS) is a structured clinical interview used to assess suicidal ideation and behavior. It includes subscales for suicidal thoughts, intent, plans, preparatory behavior, and actual suicide attempts.
  Each item is scored individually; for example:
  * Suicidal ideation severity scale: 0 (no ideation) to 5 (active ideation with specific plan and intent),
  * Behavior subscale: binary indicators (yes/no) of actual, aborted, or interrupted attempts.
  Higher scores indicate greater severity of suicide risk and behavior (i.e., a worse outcome).
Toronto Alexithymia Scale (TAS-20) | Baseline, Month 3, Month 6, Month 9, and Month 12
  The Toronto Alexithymia Scale (TAS-20) is a standardized self-report instrument designed to assess difficulties in identifying and describing emotions, and externally oriented thinking. It consists of 20 items, each rated on a 5-point Likert scale (1 = Strongly disagree to 5 = Strongly agree).
  Total scores range from 20 to 100, with higher scores indicating greater levels of alexithymia (i.e., worse emotional awareness).
Barratt Impulsiveness Scale (BIS-11) | Baseline, Month 3, Month 6, Month 9, and Month 12
  The Barratt Impulsiveness Scale - Version 11 (BIS-11) is a widely used self-report questionnaire designed to assess impulsivity as a personality trait. It consists of 30 items, rated on a 4-point Likert scale from 1 (Rarely/Never) to 4 (Almost Always/Always).
  Total scores range from 30 to 120, with higher scores indicating greater impulsivity (i.e., a worse outcome).
Difficulties in Emotion Regulation Scale - Short Form (DERS-SF) | Baseline, Month 3, Month 6, Month 9, and Month 12
  The DERS-SF (Difficulties in Emotion Regulation Scale - Short Form) is an 18-item self-report instrument that assesses difficulties in emotion regulation.
  Each item is scored on a 5-point Likert scale from 1 (Almost Never) to 5 (Almost Always). Total scores range from 18 to 90. Higher scores indicate greater difficulties in emotion regulation (i.e., a worse outcome).

SECONDARY OUTCOMES:
Rosenberg Self-Esteem Scale (RSES) | Baseline, Month 3, Month 6, Month 9, and Month 12
  The Rosenberg Self-Esteem Scale (RSES) is a widely used 10-item self-report questionnaire designed to measure global self-esteem in adolescents and adults. Each item is rated on a 4-point Likert scale (1 = Strongly Disagree to 4 = Strongly Agree), with both positively and negatively worded items.
  Total scores range from 10 to 40, with higher scores indicating higher self-esteem (i.e., a better outcome). Scores below 15 may indicate problematic low self-esteem.
Wechsler Intelligence Scale for Children (WISC-IV) / Raven's Progressive Matrices | Baseline
  Cognitive functioning is assessed at baseline using one or both of the following standardized instruments:
  * The Wechsler Intelligence Scale for Children - Fourth Edition (WISC-IV), a widely used clinical tool for measuring verbal comprehension, perceptual reasoning, working memory, and processing speed. The Full Scale IQ (FSIQ) score ranges from 40 to 160, with higher scores indicating greater cognitive ability.
  * The Raven's Progressive Matrices is a non-verbal test of abstract reasoning and fluid intelligence. Standard scores range from 60 to 140, depending on the version and age norms. Higher scores indicate higher cognitive performance.
  Only participants with IQ ≥ 80 (as determined by one of the above instruments) are included in the study.
Depression Anxiety Stress Scales - Short Version (DASS-21) | Baseline, Month 3, Month 6, Month 9, and Month 12
  The DASS-21 (Depression Anxiety Stress Scales - Short Version) is a self-report questionnaire designed to measure negative emotional states across three domains: depression, anxiety, and stress. It consists of 21 items, with 7 items per subscale. Each item is rated on a 4-point Likert scale from 0 (Did not apply to me at all) to 3 (Applied to me very much or most of the time).
  Subscale scores range from 0 to 21, and are commonly multiplied by 2 to obtain scores equivalent to the full DASS-42 (range: 0 to 42 per subscale).
  Higher scores indicate more severe symptoms (i.e., a worse outcome).)
WHO Quality of Life Questionnaire - Brief (WHOQOL-BREF) | Baseline, Month 3, Month 6, Month 9, and Month 12
  The WHOQOL-BREF is a validated, 26-item self-report questionnaire developed by the World Health Organization to assess an individual's perceived quality of life. It includes four domains:
  * Physical Health
  * Psychological Health
  * Social Relationships
  * Environment
  Each item is rated on a 5-point Likert scale, and domain scores are transformed to a scale from 0 to 100, where higher scores indicate better quality of life (i.e., a better outcome). The WHOQOL-BREF has been used across cultures and is suitable for both clinical and general populations.

OTHER OUTCOMES:
Session Rating Scale (SRS) | Each session over 10 sessions (approximately 10 weeks)
  The Session Rating Scale (SRS) is a 4-item self-report measure used to assess the therapeutic alliance at the end of each therapy session. Each item is rated on a visual analog scale from 0 to 10, yielding a total score ranging from 0 to 40.
  The four dimensions assessed are: relationship, goals and topics, approach or method, and overall alliance.
  Higher scores indicate a stronger therapeutic alliance (i.e., a better outcome). Scores below 36 may indicate a need to address ruptures in the alliance.
Outcome Rating Scale (ORS) | Each session over 10 sessions (approximately 10 weeks)
  The Outcome Rating Scale (ORS) is a 4-item self-report tool designed to measure a client's perception of change and progress in therapy. It evaluates functioning in four areas: individual (personal well-being), interpersonal (close relationships), social (work/school), and general well-being.
  Each item is scored from 0 to 10, resulting in a total score ranging from 0 to 40.
  Higher scores reflect greater perceived well-being and positive clinical change (i.e., a better outcome).

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Centro Neurolesi Bonino Pulejo, Messina, Italy, Italy